CLINICAL TRIAL: NCT04164017
Title: Comparative Evaluation of the Diagnostic Yield and Sample Quality in Endoscopic Ultrasound(EUS)-Guided Fine Needle Biopsy(FNB) of Pancreatic Solid Lesions With and Without Syringe Suction
Brief Title: Impact of Suction in the EUS-guided Fine Needle Biopsy of Solid Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Pedro Costa Moreira, Investigador Principal, Centro Hospitalar De São João, E.P.E.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 77/19
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Biopsy, Fine-Needle; Endosonography; Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided FNB with syringe suction (Experimental)
  Interventions: Device: EUS-guided FNB with Syringe Suction
- EUS-guided FNB without syringe suction (Active Comparator)
  Interventions: Device: EUS-guided FNB without Syringe Suction

INTERVENTIONS:
Device: EUS-guided FNB with Syringe Suction — For each case, FNB will be performed using two punctures: one with 20mL syringe suction and another without aspiration. The order in which they will be performed will be known only by the performing physician and the nursing team at the time that FNB is proposed. This information will be concealed from the pathologist responsible for sample analysis.
  Arms: EUS-guided FNB with syringe suction
Device: EUS-guided FNB without Syringe Suction — For each case, FNB will be performed using two punctures: one with 20mL syringe suction and another without aspiration. The order in which they will be performed will be known only by the performing physician and the nursing team at the time that FNB is proposed. This information will be concealed from the pathologist responsible for sample analysis.
  Arms: EUS-guided FNB without syringe suction

SUMMARY:
Tissue acquisition by Endoscopic Ultrasound (EUS) has become a modality of diagnosis and clinical orientation for several diseases. Although tissue acquisition traditionally involves the cytological diagnosis (using fine-needle aspiration/FNA), the importance of obtaining a core for histological examination (by fine-needle biopsy/FNB) has recently been recognized.

Currently, there is no clear establishment of the usefulness of syringe suction for the diagnostic accuracy of solid pancreatic lesions when FNB is used.

Because of that, the investigators aimed to compare sensitivity, sample adequacy, and diagnostic yield of solid pancreatic lesions EUS-guided sampling using with and without syringe suction.

The study will be conducted on a consecutive sample of patients proposed to perform EUS for solid pancreatic lesions characterization, in which the clinical and imaging findings justify the need for an FNB.

For each case, FNB will be performed using two punctures: one with 20mL syringe suction, and another without suction. The order in which they will be performed will be known only by the performing physician and the nursing team at the time that FNB is proposed. This information will be concealed from the pathologist responsible for sample analysis.

Clinical care during and after the procedure will follow the existing guidelines.

Participants will undergo a single clinical evaluation (at the time of endoscopy and recovery) without the need for follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years of age and older;
* Ability to provide free and informed consent before entering the study;
* Imaging diagnosis of a solid pancreatic lesion that was proposed for EUS characterization;
* Presence of sectional imaging method (CT/MRI) performed within six months before randomization;
* Blood test (blood count and coagulation studies) compatible with the performance of invasive maneuvers;
* Clinical indication by the endoscopist for EUS-tissue acquisition with the use of an FNB needle.

Exclusion Criteria:

* Failure to provide free and informed consent;
* Clinically significant change in haemostasis laboratory parameters: International Normalized Ratio (INR) > 1.5; activated partial thromboplastin time (aPTT)> 50 seconds; Platelets <50,000;
* Absence of a proper anticoagulant and/or anti-aggregate therapy discontinuation for the performance of FNB;
* Absence of fasting (2h without clear liquids and 6h without solid foods);
* Clinical suspicion of upper digestive tract obstruction;
* An episode of acute pancreatitis within four weeks before echoendoscopy;
* Respiratory failure or hemodynamic instability;
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield | Through study completion, an average of 10 months
  Percentage of the lesions sampled for which a tissue diagnosis is obtained and specimen adequacy is defined as the percentage of lesions sampled in which the obtained material is representative of the target site and sufficient for diagnosis
Accuracy | Through study completion, an average of 10 months
  Percentage of lesions sampled by EUS-tissue aquisition techniques that correspond to the final diagnosis at surgical histopathology or clinical follow-up (at least 12 months) for patients with nondiagnostic sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wani S, Muthusamy VR, McGrath CM, Sepulveda AR, Das A, Messersmith W, Kochman ML, Shah J. AGA White Paper: Optimizing Endoscopic Ultrasound-Guided Tissue Acquisition and Future Directions. Clin Gastroenterol Hepatol. 2018 Mar;16(3):318-327. doi: 10.1016/j.cgh.2017.10.020. Epub 2017 Oct 23. No abstract available. PMID 29074447
- [Background] Wani S, Muthusamy VR, Komanduri S. EUS-guided tissue acquisition: an evidence-based approach (with videos). Gastrointest Endosc. 2014 Dec;80(6):939-59.e7. doi: 10.1016/j.gie.2014.07.066. No abstract available. PMID 25434654
- [Background] Dwyer J, Pantanowitz L, Ohori NP, Pai RK, Vrbin C, Brand RE, Monaco SE. Endoscopic ultrasound-guided FNA and ProCore biopsy in sampling pancreatic and intra-abdominal masses. Cancer Cytopathol. 2016 Feb;124(2):110-21. doi: 10.1002/cncy.21623. Epub 2015 Oct 2. PMID 26430767
- [Background] Lee JK, Choi JH, Lee KH, Kim KM, Shin JU, Lee JK, Lee KT, Jang KT. A prospective, comparative trial to optimize sampling techniques in EUS-guided FNA of solid pancreatic masses. Gastrointest Endosc. 2013 May;77(5):745-51. doi: 10.1016/j.gie.2012.12.009. Epub 2013 Feb 21. PMID 23433878
- [Background] Wallace MB, Kennedy T, Durkalski V, Eloubeidi MA, Etamad R, Matsuda K, Lewin D, Van Velse A, Hennesey W, Hawes RH, Hoffman BJ. Randomized controlled trial of EUS-guided fine needle aspiration techniques for the detection of malignant lymphadenopathy. Gastrointest Endosc. 2001 Oct;54(4):441-7. doi: 10.1067/mge.2001.117764. PMID 11577304